CLINICAL TRIAL: NCT03682094
Title: Impact of Probiotics on Oral Microbiota in Older Adults With Dysphagia at Risk for Pneumonia
Brief Title: Impact of Probiotics on Oral Microbiota in Older Adults With Dysphagia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0428; A534255 (Other: UW Madison); SMPH/MEDICINE/GER-AD DEV (Other: UW Madison); Protocol Version 3/11/2019 (Other: UW Madison)
Record Dates: First submitted 2018-08-21; First posted 2018-09-24 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2023-07

CONDITIONS: Dysphagia
Keywords: probiotics; oral microbiome; dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Probiotics

STUDY DESIGN:
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Probiotic (Experimental): The treatment will consist of VSL#3, 3 grams (g), taken orally once a day for 4 weeks. The VSL#3 will be delivered in the form of a sachet of freeze-dried powder. Participants will be instructed to mix the sachets with water to consume. Those participants taking thickened liquids will mix the sachet with liquids thickened to the level (nectar versus honey) prescribed by their clinician. In order to facilitate delivery of the probiotic solution throughout the oral cavity, participants will be instructed to swish the solution in the mouth for up to 10 seconds (as tolerated) prior to each swallow.
  Interventions: Drug: VSL#3

INTERVENTIONS:
Drug: VSL#3 — Probiotics are dietary supplements composed of live microorganisms that are normally found within the human microbiome. Probiotics, specifically Lactobacilli and Streptococcus salivarius, have been shown to alter oral microbial composition and to inhibit oral pathogens that contribute to dental caries and periodontal disease. The probiotic chosen for this study is VSL#3, a blend of 8 strains of bacteria, including Lactobacillus and Streptococcus salivarius. VSL#3 has been well tolerated, with minimal adverse effects. VLS#3 was chosen as the treatment substance for this project due to its successful use in trials examining an array of outcomes and its combination of several strains of bacteria.
  Other Names: probiotic

SUMMARY:
The overall purpose of this study is to characterize the effect of probiotics on the oral microbiota in older adults with dysphagia at risk for pneumonia.

DETAILED DESCRIPTION:
The goal of this pilot study is to characterize the effects of probiotics on the oral microbiota in older patients with dysphagia at risk for pneumonia. A total of 20 participants will be recruited from the UW Health Inpatient Swallowing Consult Service. Participants will have a dysphagia diagnosis along with documented aspiration on videofluoroscopy. Each participant will receive a once daily VSL#3 probiotic blend (dissolved in thickened liquid as applicable) for 28 days. A baseline assessment will be completed to collect data on demographics, health history and behaviors, usual diet, level of oral intake, and patient-reported swallow function. Oral swab (buccal mucosa and tongue dorsum) as well as saliva sample collections will be completed. Data on adherence and adverse events will be collected weekly. Bacterial DNA will be extracted from oral samples and 16S rRNA sequencing techniques will be used to identify contents of oral microbiota at baseline, week 2, and week 4. Oral microbial composition will be compared between the time points, and treatment feasibility (recruitment and retention rates) in this population will be evaluated.

ELIGIBILITY:
Inclusion Criteria

1. 65 years of age or older
2. Dysphagia diagnosis based on videofluoroscopic swallow study with observed airway invasion (Penetration-Aspiration Scale score of 3 or higher)
3. Ability to provide consent
4. Ability to submit oral samples
5. Ability to swallow sachet of probiotic (dissolved in thickened liquid, as needed)
6. Ability to return to UWHC for week 2 and week 4 visits.

Exclusion Criteria

1. Currently taking antibiotics or probiotics
2. Actively receiving immunosuppressive therapy
3. Non-oral feeding with inability to swallow probiotic
4. diagnosis of head and neck cancer or upper airway disease
5. prior surgery to the head and neck region that would have affected the muscles of swallowing or the salivary glands
6. history of chemotherapy or radiation to the head and neck region
7. severe periodontal disease.
8. currently pregnant or planning to become pregnant

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Change in Oral microbiota profiles- bacterial diversity | Baseline visit, 2 weeks post-enrollment, and 4 weeks post-enrollment
  Next generation sequencing will be used to quantify the amount of alpha and beta diversity in samples collected from various locations in the oral cavity (buccal mucosa, dorsum of the tongue, saliva).

SECONDARY OUTCOMES:
Eating Assessment Test (EAT-10) | Baseline visit
  Patient reported outcome measure for swallowing
Functional Oral Intake Scale (FOIS) Score | Baseline visit
  Scale used to quantify the amount of oral versus non-oral intake
Kayser-Jones Brief Oral Health Status Examination (BOHSE) | Baseline visit
  A valid and reliable scoring instrument developed for use with older adults by non-dental health care providers.
Change in Resting Swallow Frequency Rate | Baseline visit, 2 weeks post-enrollment, and 4 weeks post-enrollment
  We will measure resting swallow frequency using surface electromyography (sEMG).
Change in Residual Mucosal Saliva (RMS) | Baseline visit, 2 weeks post-enrollment, and 4 weeks post-enrollment
  Residual Mucosal Saliva will be collected from the anterior hard palate (AHP), buccal (BUC), anterior tongue (AT), and lower labial (LL) surfaces using SialoPaper strips
Change in Amount of Saliva Produced | Baseline visit, 2 weeks post-enrollment, and 4 weeks post-enrollment
  Salivary flow rate (ml/minute) will be calculated under unstimulated and stimulated saliva collection conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States